CLINICAL TRIAL: NCT06376513
Title: Evaluation of Penile Prosthesis Pump Manipulation
Acronym: ECM3P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL24_0031
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Penile Prosthesis
Keywords: Erectile dysfunction; Penile prosthesis; Manipulation difficulties; Erection's rigidity; Sexual satisfaction
MeSH Terms: conditions — Erectile Dysfunction; Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who have undergone penile prosthesis implantation > 3 months ago and their partner (Other): Evaluation of the manipulation abilities of patients with penile prostheses Evaluation of the rigidity of erections with penile prosthesis, the patient and partner's sexual satisfaction, the satisfaction related to pump manipulation
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Evaluation of the manipulation abilities of patients with penile prostheses Evaluation of the rigidity of erections with penile prosthesis, the patient and partner's sexual satisfaction, the satisfaction related to pump manipulation

SUMMARY:
Erectile dysfunction is a highly prevalent pathology. When oral or injectable pharmacological treatments prove ineffective, the treatment of choice is penile prosthesis which provides the possibility of sexual activity with penetration.

Unfortunately, current prostheses are difficult (or even impossible) to manipulate for some patients. Many patients underutilize their device due to difficulties in using the pump related to mechanical issues (difficult grip, lack of strength, etc.) or sensory issues (altered proprioception, etc.), resulting in an inability to achieve rigidity that allows optimal satisfaction for the patient and/or partners.

These difficulties correspond to a significant portion of dissatisfaction among patients with penile prostheses.

Actually, no study has evaluated patients' ability to manipulate the pump of their penile prosthesis, as well as the association between these manipulation abilities, the rigidity of erections with a penile prosthesis, and patient and partner sexual satisfaction.

In this descriptive study, the primary outcome is to describe the manipulation abilities of patients with penile prostheses during follow-up consultations after prosthesis implantation.

The secondary outcomes are to estimate the association of various markers related to penile prosthesis manipulation (overall hand grip strength, pinch grip strength, proprioception, and discrimination) with

* Rigidity of erections with penile prosthesis
* Patient's sexual satisfaction
* Partner's sexual satisfaction
* Satisfaction related to pump manipulation

ELIGIBILITY:
Inclusion Criteria:

* The patients will be included based on the following criteria:
* Adults
* Erectile Dysfunction, and had undergone penile prosthesis implantation for more than 3 months
* Able to comprehend the nature and purpose of the research
* Having provided informed consent

The partner will be included based on the following criteria :

* Adults
* Having a partner who meets the inclusion criteria
* Able to comprehend the nature and purpose of the research
* Having provided informed consent

Exclusion Criteria:

* Patients with a dysfunctional penile prosthesis (reservoir, pump, or cylinders anomaly)
* Adults subject to legal protective measures.
* Individuals not affiliated with a social security scheme or beneficiaries of a similar scheme.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with penile prosthesis
Enrollment: 60 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Describing the manipulation abilities of patients with penile prosthesis : overall hand grip strength | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  Measurement of overall hand grip strength using the JAMAR dynamometer. The force is expressed in kg.
Describing the manipulation abilities of patients with penile prosthesis : pinch grip strength | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  Measurement of pinch grip strength using the "pinch test".The force is expressed in kg.
Describing the manipulation abilities of patients with penile prosthesis : proprioception | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  Measurement of proprioception with a object recognition test : the "Moberg pick-up test".
  The patient must recognize (with eyes closed) objects that he has previously seen and held in his hand. A score ranging from 0 to 12 will thus be obtained.
Describing the manipulation abilities of patients with penile prosthesis :discrimination | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  Measurement of discrimination with a two points touch test. Evaluation of the smallest perceived distance between two points, expressed in mm.
Describing the manipulation abilities of patients with penile prosthesis :upper limb function for activities of daily living | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  Evaluation of upper limb function for activities of daily living: the Quick DASH (Disabilities of the Arm, Shoulder and Hand).
  A score ranging from 11 to 55 will thus be obtained.

SECONDARY OUTCOMES:
Correlation of manipulation parameters (main outcome) with rigidity of erections | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  estimate the association of various markers related to penile prosthesis manipulation (overall hand grip strength, pinch grip strength, proprioception, and discrimination) with rigidity of erections with penile prosthesis.
  The patient will be asked to inflate his prosthesis under normal usage conditions. The physician will then apply the device to the erect penis and note the point of deformation of the penis (buckling). The result is expressed in grams.
  Manipulation of the penile prosthesis pump resulting in an erection rigidity exceeding 550g will be considered adequate
Correlation of manipulation parameters (main outcome) with patient's sexual satisfaction modified EDITS | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  To estimate the association of various markers related to penile prosthesis manipulation (overall hand grip strength, pinch grip strength, proprioception, and discrimination) with patient's sexual satisfaction (modified EDITS).
  The responses to the EDITS questionnaire are given on a Likert scale ranging from 0 to 4 for each item. A score of 0 corresponds to maximum dissatisfaction, and a score of 4 corresponds to maximum satisfaction. A score ranging from 0 to 36 will thus be obtained. For each item, satisfaction is deemed sufficient if the Likert score obtained is ≥ 3.
Correlation of manipulation parameters (main outcome) with patient's sexual satisfaction QoLSPP | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  To estimate the association of various markers related to penile prosthesis manipulation (overall hand grip strength, pinch grip strength, proprioception, and discrimination) with patient's sexual satisfaction ( QoLSPP).
  The responses to the QoLSPP questionnaire are given on a Likert scale ranging from 0 to 5 for each item. A score of 0 corresponds to maximum dissatisfaction, and a score of 5 corresponds to maximum satisfaction. A score ranging from 0 to 80 will thus be obtained. For each item, satisfaction is deemed sufficient if the Likert score obtained is ≥ 3.
Correlation of manipulation parameters (main outcome) with partner's sexual satisfaction | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  To estimate the association of various markers related to penile prosthesis manipulation (overall hand grip strength, pinch grip strength, proprioception, and discrimination) with partner's sexual satisfaction (partner modified EDITS)
  The responses to the partner EDITS questionnaire are given on a Likert scale ranging from 0 to 4 for each item. A score of 0 corresponds to maximum dissatisfaction, and a score of 4 corresponds to maximum satisfaction. A score ranging from 0 to 20 will thus be obtained. For each item, satisfaction is deemed sufficient if the Likert score obtained is ≥ 3.
Correlation of manipulation parameters (main outcome) with satisfaction related to pump manipulation (self-made questionnaire) | At inclusion (during a standard of care follow-up consultation from 3 months post-surgery)
  To estimate the association of various markers related to penile prosthesis manipulation (overall hand grip strength, pinch grip strength, proprioception, and discrimination) with satisfaction related to pump manipulation (self-made questionnaire)
  The responses to this questionnaire will also be provided on a Likert scale ranging from 0 to 4 for each item. A score of 0 corresponds to complete inability to perform the act, and a score of 4 corresponds to performing the act without any difficulty. A score ranging from 0 to 24 will thus be obtained. For each item, satisfaction related to pump manipulation is deemed sufficient if the Likert score obtained is ≥ 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Lyon Sud Hospital,, Pierre-Bénite, France